CLINICAL TRIAL: NCT00005235
Title: The Ability of Several Short-term Measures of RR Variability to Predict Mortality After Myocardial Infarction
Brief Title: Heart Rate Variability and Sudden Cardiac Death
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CUMC ID unknown (1116); R01HL041552 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Death, Sudden, Cardiac; Ventricular Arrhythmia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the ability of heart rate variability to identify myocardial infarction patients at high risk of dying, particularly from sudden cardiac death.

DETAILED DESCRIPTION:
BACKGROUND:

Sudden cardiac death usually is caused by malignant ventricular arrhythmias. Malignant ventricular arrhythmias in coronary heart disease are due to an interplay among substrate such as scarred ventricles, triggering events such as spontaneous ventricular arrhythmias, and the autonomic nervous system. Non-invasive methods were needed to evaluate these three components of risk in order to develop comprehensive detection and prevention programs. Non-invasive screening tests for the arrhythmogenic substrate include left ventricular ejection fraction and signal-averaged electrocardiograms, and for triggering events, the 24-hour continuous ECG recordings. Measures of heart rate variability defined as the variability of the instantaneous heart rates or heart period variability defined as variability of the normal R-R intervals may provide the means for non-invasive assessment of autonomic nervous system activity. In previous studies it has been shown that a broad band measure of heart period variability, the standard deviation of all normal R-R intervals in a continuous 24-hour ECG recording made eight to fourteen days after myocardial infarction, predicted mortality in the subsequent two to four years independently of left ventricular dysfunction and spontaneous ventricular arrhythmias.

The six multicenter studies from which the data were drawn included: the Multicenter Post Infarction Program (MPIP), a longitudinal, observational study of 867 patients; the Multicenter Diltiazem Post Infarction Trial (MDPIT), a double-blind, randomized, placebo-controlled trial of 2,466 patients; the Cardiac Arrhythmia Pilot Study (CAPS), a double-blind, randomized, placebo-controlled trial of 502 patients; the Cardiac Arrhythmia Suppression Trial (CAST), a double-blind, randomized, placebo-controlled trial of 4,200 patients; Electrophysiologic Studies Versus Electrocardiographic Monitoring (ESVEM), a comparison of two methods for evaluating antiarrhythmic drug efficacy in 350 patients; and the Cardiac Rate/Rhythm in Normal Adults, a cross-sectional observational study of 250 subjects.

DESIGN NARRATIVE:

Measurements of short and long-term heart rate and heart period variability were compared. The day-to-day reproducibility and time course of change were determined in measures of heart rate variability and heart period variability in patients with myocardial infarction. The predictive accuracy of heart rate variability measured late after myocardial infarction for subsequent mortality and development of malignant ventricular arrhythmias was determined. Heart rate and heart period variability findings after myocardial infarction were compared with those in age and sex-matched normal subjects and with those made in patients with malignant ventricular arrhythmias.

ELIGIBILITY:
Inclusion criteria

--Patients that have had myocardial infarction within 2 weeks - still in hospital and sedentary except for short walks in hospital corridors

Exclusion criteria

--Inadequate 24-hour ECG recordings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in the Multicenter Post Infarction Program (MPIP), a natural history study
Sampling Method: Non-Probability Sample
Enrollment: 715 (Actual)
Dates: Start 1988-12; Primary Completion 1993-09 (Actual); Study Completion 1993-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Bigger, MD, Principal Investigator — Professor Emeritus of Medicine and Pharmacology, Columbia University
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Background] Bigger JT Jr, Albrecht P, Steinman RC, Rolnitzky LM, Fleiss JL, Cohen RJ. Comparison of time- and frequency domain-based measures of cardiac parasympathetic activity in Holter recordings after myocardial infarction. Am J Cardiol. 1989 Sep 1;64(8):536-8. doi: 10.1016/0002-9149(89)90436-0. No abstract available. PMID 2773799
- [Background] Bigger JT Jr, La Rovere MT, Steinman RC, Fleiss JL, Rottman JN, Rolnitzky LM, Schwartz PJ. Comparison of baroreflex sensitivity and heart period variability after myocardial infarction. J Am Coll Cardiol. 1989 Nov 15;14(6):1511-8. doi: 10.1016/0735-1097(89)90390-2. PMID 2809012
- [Background] Rottman JN, Steinman RC, Albrecht P, Bigger JT Jr, Rolnitzky LM, Fleiss JL. Efficient estimation of the heart period power spectrum suitable for physiologic or pharmacologic studies. Am J Cardiol. 1990 Dec 15;66(20):1522-4. doi: 10.1016/0002-9149(90)90551-b. No abstract available. PMID 2252008
- [Background] Bigger JT Jr, Fleiss JL. The variability of spontaneous ventricular arrhythmias in the year after myocardial infarction. J Am Coll Cardiol. 1991 Jan;17(1):9-10. doi: 10.1016/0735-1097(91)90698-9. No abstract available. PMID 1702796
- [Background] Goldsmith RL, Bigger JT Jr, Steinman RC, Fleiss JL. Comparison of 24-hour parasympathetic activity in endurance-trained and untrained young men. J Am Coll Cardiol. 1992 Sep;20(3):552-8. doi: 10.1016/0735-1097(92)90007-a. PMID 1512332
- [Background] Fleiss JL, Bigger JT Jr, Rolnitzky LM. The correlation between heart period variability and mean period length. Stat Med. 1992 Jan 15;11(1):125-9. doi: 10.1002/sim.4780110111. PMID 1557568
- [Background] Bigger JT Jr, Fleiss JL, Steinman RC, Rolnitzky LM, Kleiger RE, Rottman JN. Correlations among time and frequency domain measures of heart period variability two weeks after acute myocardial infarction. Am J Cardiol. 1992 Apr 1;69(9):891-8. doi: 10.1016/0002-9149(92)90788-z. PMID 1550018
- [Background] Bigger JT Jr, Fleiss JL, Rolnitzky LM, Steinman RC. Stability over time of heart period variability in patients with previous myocardial infarction and ventricular arrhythmias. The CAPS and ESVEM investigators. Am J Cardiol. 1992 Mar 15;69(8):718-23. doi: 10.1016/0002-9149(92)90493-i. PMID 1546643
- [Background] Bigger JT Jr, Fleiss JL, Steinman RC, Rolnitzky LM, Kleiger RE, Rottman JN. Frequency domain measures of heart period variability and mortality after myocardial infarction. Circulation. 1992 Jan;85(1):164-71. doi: 10.1161/01.cir.85.1.164. PMID 1728446
- [Background] Bigger JT Jr, Fleiss JL, Rolnitzky LM, Steinman RC, Schneider WJ. Time course of recovery of heart period variability after myocardial infarction. J Am Coll Cardiol. 1991 Dec;18(7):1643-9. doi: 10.1016/0735-1097(91)90497-w. PMID 1960309
- [Background] Kleiger RE, Bigger JT, Bosner MS, Chung MK, Cook JR, Rolnitzky LM, Steinman R, Fleiss JL. Stability over time of variables measuring heart rate variability in normal subjects. Am J Cardiol. 1991 Sep 1;68(6):626-30. doi: 10.1016/0002-9149(91)90355-o. PMID 1877480
- [Background] Cook JR, Bigger JT Jr, Kleiger RE, Fleiss JL, Steinman RC, Rolnitzky LM. Effect of atenolol and diltiazem on heart period variability in normal persons. J Am Coll Cardiol. 1991 Feb;17(2):480-4. doi: 10.1016/s0735-1097(10)80119-6. PMID 1991906
- [Background] Bigger JT Jr, Rolnitzky LM, Steinman RC, Fleiss JL. Predicting mortality after myocardial infarction from the response of RR variability to antiarrhythmic drug therapy. J Am Coll Cardiol. 1994 Mar 1;23(3):733-40. doi: 10.1016/0735-1097(94)90761-7. PMID 7509355
- [Background] Bloomfield DM, Bigger JT Jr, Pavri BB, Han J, Fleiss JL, Rolnitzky LM, Steinman RC. Vagal modulation of RR intervals during head-up tilt and the infusion of isoproterenol. Am J Cardiol. 1995 Jun 1;75(16):1145-50. doi: 10.1016/s0002-9149(99)80747-4. PMID 7762502
- [Background] Bigger JT Jr, Fleiss JL, Steinman RC, Rolnitzky LM, Schneider WJ, Stein PK. RR variability in healthy, middle-aged persons compared with patients with chronic coronary heart disease or recent acute myocardial infarction. Circulation. 1995 Apr 1;91(7):1936-43. doi: 10.1161/01.cir.91.7.1936. PMID 7895350
- [Background] Bigger JT, Fleiss JL, Rolnitzky LM, Steinman RC. The ability of several short-term measures of RR variability to predict mortality after myocardial infarction. Circulation. 1993 Sep;88(3):927-34. doi: 10.1161/01.cir.88.3.927. PMID 8353919
- [Background] Kaufman ES, Bosner MS, Bigger JT Jr, Stein PK, Kleiger RE, Rolnitzky LM, Steinman RC, Fleiss JL. Effects of digoxin and enalapril on heart period variability and response to head-up tilt in normal subjects. Am J Cardiol. 1993 Jul 1;72(1):95-9. doi: 10.1016/0002-9149(93)90226-3. PMID 8517437
- [Background] Bigger JT Jr, Fleiss JL, Rolnitzky LM, Steinman RC. Frequency domain measures of heart period variability to assess risk late after myocardial infarction. J Am Coll Cardiol. 1993 Mar 1;21(3):729-36. doi: 10.1016/0735-1097(93)90106-b. PMID 8436755
- Available data/document: NCBI website — http://www.ncbi.nlm.nih.gov/pubmed/8353919